CLINICAL TRIAL: NCT00376298
Title: Urology Database for Outcomes Research
Brief Title: Urology Database to Evaluate Clinical Information and Improve Patient Care.
Status: Completed | Type: Observational
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2004-050
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Incontinence; Prostate Cancer; Interstitial Cystitis; Urinary Retention; Pelvic Organ Prolapse
Keywords: incontinence; prostate cancer; interstitial cystitis
MeSH Terms: conditions — Prostatic Neoplasms; Cystitis, Interstitial; Urinary Retention; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of initiating the Urology Database is to evaluate the outcomes of urology procedures and medical management to enhance the care and treatment of urology patients.

DETAILED DESCRIPTION:
The current study population will include all patients having had a radical prostatectomy for the treatment of prostate cancer, surgical prolapse repair as well as patients having had InterStim sacral nerve stimulator implantation. The database will house data extracted from the medical records. Patient demographics, and preoperative, intra-operative, postoperative, and follow-up clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing radical prostatectomy, pelvic organ prolapse repair and neurostimulator (Interstim) implantation at William Beaumont Hospital beginning January 1, 1998, as well as other urology patients as research questions are identified. Only patients who have accepted William Beaumont Hospital's Privacy Notices will be included in the database.

Exclusion Criteria:

Patients not acknowledging acceptance of William Beaumont Hospital's Privacy Notices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and Women with conditions including radical prostatectomy, pelvic organ prolapse and neurostimulator implantation at William Beaumont Hospital
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2004-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States